CLINICAL TRIAL: NCT05040295
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, CROSS-OVER, SINGLE DOSE STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF PEDIATRIC RITLECITINIB (PF-06651600) CAPSULES AND SPRAY CONGEALED BEADS RELATIVE TO ADULT CAPSULES IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Single Dose Study To Test Two Pediatric Forms Of Ritlecitinib Compared With Adult Ritlecitinib In Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981030
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Results first posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence 1 (Experimental): Treatment sequence 1 will receive a single 30 milligrams (mg) ritlecitinib intact adult capsule during the first period, three 10 mg ritlecitinib pediatric capsules during the second period and 30 mg ritlecitinib spray congealed beads in the third period.
  Interventions: Drug: ritlecitinib
- Treatment Sequence 2 (Experimental): Treatment sequence 2 will receive three 10 mg ritlecitinib pediatric capsules during the first period, a single 30 mg intact adult capsule during the second period and 30 mg ritlecitinib spray congealed beads in the third period.
  Interventions: Drug: ritlecitinib

INTERVENTIONS:
Drug: ritlecitinib — 30 mg intact adult capsule
Drug: ritlecitinib — 10 mg pediatric capsule
Drug: ritlecitinib — 30 mg spray congealed beads

SUMMARY:
A phase I, single dose study to test two forms of pediatric ritlecitinib compared to adult ritlecitinib in healthy adults aged 18-55 years old. Approximately 12 adults will participate for approximately 2.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by medical evaluation including a detailed medical history, complete (full) physical examination, which includes BP and pulse rate measurement, clinical laboratory tests, and 12-lead ECG.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Known immunodeficiency disorder, including positive serology for HIV at screening, or a first degree relative with a hereditary immunodeficiency
* Infection with hepatitis B or hepatitis C viruses.
* History of any lymphoproliferative disorder
* Known present or a history of malignancy other than a successfully treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Saadeddin A, Purohit V, Huh Y, Wong M, Maulny A, Dowty ME, Sagawa K. Virtual Bioequivalence Assessment of Ritlecitinib Capsules with Incorporation of Observed Clinical Variability Using a Physiologically Based Pharmacokinetic Model. AAPS J. 2024 Jan 24;26(1):17. doi: 10.1208/s12248-024-00888-9. PMID 38267790
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981030

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 participants were assigned to study treatment and all the participants were treated in this study.
Groups:
- [Sequence 1] Ritlecitinib: Intact Adult Capsule=>Pediatric Capsules=>Spray Congealed Beads: Participants underwent 3 periods and received a single dose of study drug in each period. Participants received ritlecitinib 30 mg intact adult capsule single dose (SD) on Period 1 Day 1, followed by ritlecitinib 3*10 mg pediatric capsules SD on Period 2 Day 1, and ritlecitinib 30 mg spray congealed beads SD on Period 3 Day 1. There was a at least 2-day washout between dosing.
- [Sequence 2] Ritlecitinib: Pediatric Capsules=>Intact Adult Capsule=>Spray Congealed Beads: Participants underwent 3 periods and received a single dose of study drug in each period. Participants received ritlecitinib 3*10 mg pediatric capsules SD on Period 1 Day 1, followed by ritlecitinib 30 mg intact adult capsule SD on Period 2 Day 1, and ritlecitinib spray congealed beads 30 mg on Period 3 Day 1. There was a at least 2-day washout between dosing.
Period: Period 1
Arm/Group | [Sequence 1] Ritlecitinib: Intact Adult Capsule=>Pediatric Capsules=>Spray Congealed Beads | [Sequence 2] Ritlecitinib: Pediatric Capsules=>Intact Adult Capsule=>Spray Congealed Beads
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | [Sequence 1] Ritlecitinib: Intact Adult Capsule=>Pediatric Capsules=>Spray Congealed Beads | [Sequence 2] Ritlecitinib: Pediatric Capsules=>Intact Adult Capsule=>Spray Congealed Beads
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 3
Arm/Group | [Sequence 1] Ritlecitinib: Intact Adult Capsule=>Pediatric Capsules=>Spray Congealed Beads | [Sequence 2] Ritlecitinib: Pediatric Capsules=>Intact Adult Capsule=>Spray Congealed Beads
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Entire Study Population: Includes all participants who were assigned to study treatment. Participants assigned to treatment sequence 1 received ritlecitinib 30 mg intact adult capsule SD on Period 1 Day 1, followed by ritlecitinib 3*10 mg pediatric capsules SD on Period 2 Day 1, and ritlecitinib 30 mg spray congealed beads SD on Period 3 Day 1. Participants assigned to treatment sequence 2 received ritlecitinib 3*10 mg pediatric capsules SD on Period 1 Day 1, followed by ritlecitinib 30 mg intact adult capsule SD on Period 2 Day 1, and ritlecitinib 30 mg spray congealed beads SD on Period 3 Day 1. There was a at least 2-day washout between dosing.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: Years] | 40.0 [23 to 56]
Age, Customized [Count of Participants; unit: Participants]
  18-44 Years | 8
  45-64 Years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5
  Black or African American | 3
  Asian | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) for Ritlecitinib
Description: Plasma AUCinf for ritlecitinib is reported. AUCinf was calculated as [AUClast+(Clast*/kel)], where AUClast is the area under the plasma concentration-time profile from time 0 to the time of the Clast, Clast is the last quantifiable concentration, Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, and 24 hours post dose on Day 1 in each period
Population: Includes all participants randomized and treated who had at least 1 of the pharmacokinetic (PK) parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Groups:
- Treatment A: Ritlecitinib 30 mg Intact Adult Capsule: Participants who were assigned to Treatment sequence 1 received a single dose of ritlecitinib 30 mg intact adult capsule on Period 1 Day 1. Participants who were assigned to Treatment sequence 2 received a single dose of ritlecitinib 30 mg intact adult capsule on Period 2 Day 1.
- Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules: Participants who were assigned to Treatment sequence 1 received a single dose of ritlecitinib 3*10 mg pediatric capsules on Period 2 Day 1. Participants who were assigned to Treatment sequence 2 received a single dose of ritlecitinib 3*10 mg pediatric capsules on Period 1 Day 1.
- Treatment C: Ritlecitinib 30 mg Spray Congealed Beads: Participants received a single dose of ritlecitinib 30 mg spray congealed beads on Period 3 Day 1.
Arm/Group | Treatment A: Ritlecitinib 30 mg Intact Adult Capsule | Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules | Treatment C: Ritlecitinib 30 mg Spray Congealed Beads
Number analyzed (Participants) | 12 | 12 | 12
nanograms*hours/milliliter (ng*hr/mL) | 361.1 (39) | 370.1 (40) | 385.1 (38)
Statistical Analysis 1: Comparison: Treatment A: Ritlecitinib 30 mg Intact Adult Capsule vs Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules; AUCinf was analyzed using a mixed effects model with sequence and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model; Test type: Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Ratio of adjust geometric means = 102.50, 90% CI 2-sided [94.21 to 111.51] — Reference = Treatment A Test = Treatment B Ratio=Test/Reference
Statistical Analysis 2: Comparison: Treatment A: Ritlecitinib 30 mg Intact Adult Capsule vs Treatment C: Ritlecitinib 30 mg Spray Congealed Beads; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjust geometric means = 106.65, 90% CI 2-sided [100.07 to 113.66] — Reference = Treatment A Test = Treatment C Ratio=Test/Reference

2. Primary Outcome: Maximum Plasma Concentration (Cmax) for Ritlecitinib
Description: Plasma Cmax for ritlecitinib is reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 16, and 24 hours post dose on Day 1 in each period
Population: Includes all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A: Ritlecitinib 30 mg Intact Adult Capsule | Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules | Treatment C: Ritlecitinib 30 mg Spray Congealed Beads
Number analyzed (Participants) | 12 | 12 | 12
ng/mL | 197.4 (38) | 199.6 (37) | 177.9 (30)
Statistical Analysis 1: Comparison: Treatment A: Ritlecitinib 30 mg Intact Adult Capsule vs Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules; Cmax was analyzed using a mixed effects model with sequence and treatment as fixed effects and participant within sequence as a random effect. Estimates of the adjusted mean differences (Test-Reference) and corresponding 90% confidence intervals (CIs) were obtained from the model; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjust geometric means = 101.12, 90% CI 2-sided [88.25 to 115.87] — Reference = Treatment A Test = Treatment B Ratio=Test/Reference
Statistical Analysis 2: Comparison: Treatment A: Ritlecitinib 30 mg Intact Adult Capsule vs Treatment C: Ritlecitinib 30 mg Spray Congealed Beads; [analysis description as in outcome 2, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of adjust geometric means = 90.11, 90% CI 2-sided [78.49 to 103.44] — Reference = Treatment A Test = Treatment C Ratio=Test/Reference

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (All Causalities and Treatment-Related)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Treatment-emergent AEs (TEAEs) = between first dose of study treatment and up to 35 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-related AEs and SAEs were determined by the investigator. Severe=an event that prevents normal everyday activities.
Time Frame: Post first dose of study intervention on Period 1 Day 1 up to 35 days post last dose of study intervention on Period 3 Day 1 (maximum of 40 days)
Population: Includes all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Ritlecitinib 30 mg Intact Adult Capsule | Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules | Treatment C: Ritlecitinib 30 mg Spray Congealed Beads
Number analyzed (Participants) | 12 | 12 | 12
Participants
  Participants with AEs (All Causalities) | 2 | 1 | 1
  Participants with AEs (Treatment Related) | 0 | 0 | 0
  Participants with SAEs | 0 | 0 | 0
  Participants with Severe AEs | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline Abnormality
Description: Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes, etc), chemistry (fasting glucose, calcium, sodium, potassium, chloride, total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, uric acid, total protein, albumin, etc), and urinalysis (glucose, protein, blood, ketones, nitrites, leukocyte esterase, etc). Baseline = the last pre-dose measurement before Period 1 Day 1 (ie, first dose of study intervention). Laboratory abnormalities meeting pre-defined criteria are reported for this outcome measure. ULN=upper limit of normal. LLN=lower limit of normal. HPF=high-powered field. mEq=milliequivalent. L=liter.
Time Frame: Baseline up to Period 3 Day 2 (maximum of 7 days)
Population: Includes all participants assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Participants
  Eosinophils/Leukocytes (%) >1.2*ULN | 1
  Monocytes/Leukocytes (%) >1.2*ULN | 2
  Bicarbonate (mEq/L) <0.9*LLN | 1
  Ketones (No Unit) >=1 | 1
  URINE Hemoglobin (No Unit) >=1 | 1
  Nitrite (No Unit) >=1 | 1
  Leukocyte Esterase (No Unit) >=1 | 1
  URINE Leukocytes (/HPF) >=20 | 1
  Bacteria (/HPF) >20 | 1

ADVERSE EVENTS:
Time Frame: Baseline (ie, post the first dose of study intervention) up to 35 days post last dose of study intervention (maximum of 40 days)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Treatment A: Ritlecitinib 30 mg Intact Adult Capsule | Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules | Treatment C: Ritlecitinib 30 mg Spray Congealed Beads
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Ritlecitinib 30 mg Intact Adult Capsule (N=12) | Treatment B: Ritlecitinib 3*10 mg Pediatric Capsules (N=12) | Treatment C: Ritlecitinib 30 mg Spray Congealed Beads (N=12)
Fatigue (General disorders) | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT05040295/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT05040295/SAP_001.pdf